CLINICAL TRIAL: NCT03859791
Title: "True Incidence of Hip Dislocation After Primary THA - a Nationwide Population Study"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Lars Lykke Hermansen, MD, Ph.d. Student, University of Southern Denmark
Other Study IDs: 3-3013-2128/1
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Hip Dislocation
MeSH Terms: conditions — Hip Dislocation | interventions — Tacrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: THA — Study participants have received a total hip arthroplasty due to arthritis. We do not make further intervention.

SUMMARY:
The primary objective is to report the true incidence of hip dislocations in primary THA patients within 2 years of index surgery.

Secondary, patient and component characteristics (age, sex, comorbidity, cemented/uncemented, approach, head diameter) are analyzed as potential risk factors for dislocation. Specific components may be analyzed based on number.

DETAILED DESCRIPTION:
Based on published literature and personal experience, most hip surgeons have an assumption of the degree of hip dislocation. This will be the first study to reveal the actual extent of this specific complication in a large population. It will give surgeons knowledge of the current standards -both on a national and hospital level. Depending on the results and comparisons to relevant countries, the investigators will be able to either substantiate or forced to rethink current procedures. This applies to both surgical access and use of specific components.

Since the vast majority of dislocations appear within 1-2 years after primary surgery (29), the follow-up period will be 2 years. By applying the National Patient Registry the investigators are able to identify any type of patient contact with the hospital system throughout Denmark in these 2 years. Patients assigned with correct diagnostic and procedural codes for dislocation and reduction are identified. However, the investigators will also find the cases of dislocation that are incorrectly coded in the registry. Therefore, the investigators will manually look in all the patient files from orthopedic contacts regardless of assigned diagnostic and procedural codes. Additionally, emergency room and internal medicine contacts are scanned with a broad and comprehensive range of relevant hip- and dislocation-related codes to identify episodes of hip dislocation, which are incorrectly coded. These patient files will also be manually reviewed.

If a patient is revised within the first 2 years, the follow-up period ends on the revision date. Revisions are also registered in the Danish Hip Arthroplasty Registry. However, the completeness is 93-95% and therefore lower than for primary operations. In order to have the complete set of revisions, the investigators will enrich our data with an extraction from the National Patient Registry by applying all approved hip revision codes

ELIGIBILITY:
Inclusion Criteria:

* patients with the diagnosis "primary/idiopathic hip OA and inserted THA from 01.01.2010 - 31.12.2014.

Exclusion Criteria:

* patients receiving a resurfacing hip arthroplasty and hip revisions
* patients with incomplete registry data
* patients with previous hip surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective, we include patients with the diagnosis "primary/idiopathic hip OA". Patients are identified by data extraction from the Danish Hip Arthroplasty Registry. From 2010-2014 an average of 9000 hips/year received a primary THA and about 80% of these patients were diagnosed with idiopathic/primary arthritis. Therefore, we tend to include approximately 36.000 hips. We also include the second hip, if a patient undergoes 2 primary operations in our inclusion period and this is adjusted for in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 32500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Hip dislocation | 2 years.
  The true incidence of hip dislocation calculated as proportion presented with 95% confidence intervals (CI).

SECONDARY OUTCOMES:
Age | 2 years.
  Potential risk factor found by logistic regression analysis
Sex | 2 years.
  Potential risk factor found by logistic regression analysis
Comorbidity | 2 years.
  Potential risk factor found by logistic regression analysis
Fixation of components | 2 years.
  Potential risk factor found by logistic regression analysis
Surgical approach | 2 years.
  Potential risk factor found by logistic regression analysis
Head diameter of prosthesis | 2 years.
  Potential risk factor found by logistic regression analysis
Time to dislocation | 2 years.
  Time to first dislocation presented by Kaplan-Meier plot.
Development in complication (dislocation) over time. | 5 years.
  Incidence each year (2010-2014) calculated as proportion presented with 95% confidence intervals (CI) and compared statistically depending on distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of South West Jutland, Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.